CLINICAL TRIAL: NCT02979171
Title: Comparison in Difficult Airway Scenario Induced in Patients With Laryngeal Mask Airway (LMA)-Classic™, LMA™ - Flexible and LMA - Proseal™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 71146310
Record Dates: First submitted 2016-04-05; First posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Difficult Airway

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- LMA-Classic (Active Comparator): airway management with LMA-Classic
  Interventions: Device: Laryngeal Mask Airway Classic
- LMA-Flexible (Active Comparator): airway management with LMA-Flexible
  Interventions: Device: Laryngeal Mask Airway Classic
- LMA-Proseal (Active Comparator): airway management with LMA-Proseal
  Interventions: Device: Laryngeal Mask Airway Classic

INTERVENTIONS:
Device: Laryngeal Mask Airway Classic

SUMMARY:
Supraglottic airway tools, one of the tools used in the management of the difficult airway. American Society of Anesthesiologists and the Difficult Airway Society of the United Kingdom airway management algorithms have included the LMA. In our study investigators aimed to determine which one will show the best performance with supraglottic airway means that LMA - Classic, LMA - Flexible and LMA - ProSeal in patients that difficult airway scenarios created with attaching collar.

ELIGIBILITY:
Inclusion Criteria:

* Without a history of difficult intubation, supine position, does not require tracheal intubation, undergo elective surgery

Exclusion Criteria:

* High aspiration risk, who take more than 4 hours surgery
* Body mass index greater than of 35 kg/m²
* Disease related to the cervical spine
* The mouth opening is less than 20 mm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
insertion time and attempts in min. | through study completion, an average of 6 months
oropharyngeal leak pressure in cmH20. | through study completion, an average of 6 months
fiberoptic view grade by Brimacombe and Berry bronchoscopy score | through study completion, an average of 6 months
  score1-4 (easy to difficult)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Science University, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided